CLINICAL TRIAL: NCT06891105
Title: Effect of Probiotic and Synbiotic Administration on the Nutritional Status of Hemodialysis Patients. a Randomized Controlled Trial
Brief Title: Effect of Probiotic and Synbiotic Administration on Nutritional Status in Hemodialysis Patients
Acronym: ProSyn-HD
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Walaa Mamdouh Mohamed Mahmoud, Principal Investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS.23.05.2418
Record Dates: First submitted 2025-03-18; First posted 2025-03-24 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Hemodialysis; Probiotics; Synbiotics; Nutritional Status
Keywords: End-Stage Renal Disease; Hemodialysis; Probiotics; Synbiotics; Nutritional Status; Gut Microbiota
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (No Intervention) (No Intervention): This arm will include 20 participants who will not receive any treatment. The purpose of this group is to serve as a baseline for comparison with the two intervention arms. Participants will undergo regular hemodialysis treatment, but no probiotic or synbiotic supplementation will be provided.
- Probiotic Group (Experimental): This arm will consist of 20 participants who will receive daily probiotic supplementation (Lactogemikan from Pescado Company, containing Lactobacillus plantarum). The objective is to evaluate the effect of probiotics on the nutritional status, including BMI, skin fold thickness, and protein metabolism in hemodialysis patients. Participants will receive the probiotic for a duration of 6 months.
  Interventions: Dietary Supplement: Lactogemikan (Probiotic Supplement)
- Synbiotic Group (Experimental): This arm will include 20 participants who will receive daily synbiotic supplementation, which includes both probiotics (Lactogemikan from Pescado Company) and prebiotic fiber (oat, 3g/day). The purpose of this arm is to assess the impact of synbiotics on the nutritional status and gut microbiota balance of hemodialysis patients. Participants will receive the synbiotic for 6 months.
  Interventions: Dietary Supplement: Lactogemikan + Prebiotic Fiber (Synbiotic Supplement)

INTERVENTIONS:
Dietary Supplement: Lactogemikan (Probiotic Supplement) — This intervention involves daily supplementation of Lactogemikan from Pescado Company, which contains Lactobacillus plantarum, a well-known probiotic strain. The probiotic is intended to improve gut microbiota balance, which may lead to improved nutritional status and health outcomes in hemodialysis patients. The dosage is one tablet daily for a duration of six months.
  Arms: Probiotic Group
Dietary Supplement: Lactogemikan + Prebiotic Fiber (Synbiotic Supplement) — This intervention involves daily supplementation of Lactogemikan (containing Lactobacillus plantarum) combined with prebiotic fibers from oat (3g per day). The synbiotic is designed to provide the benefits of both probiotics (to balance gut microbiota) and prebiotics (to support the growth of beneficial bacteria). This intervention is intended to improve the nutritional status of hemodialysis patients over a 6-month period. The dosage is one tablet daily, combined with 3g of oat fiber.
  Arms: Synbiotic Group

SUMMARY:
This study aims to investigate the impact of probiotics and synbiotics on the nutritional status of patients with end-stage kidney disease (ESRD) who are undergoing hemodialysis. ESRD patients often face challenges such as poor nutritional status, increased risk of infections, and imbalances in gut microbiota. These challenges are made worse by the frequent use of medications, dietary restrictions, and the hemodialysis process itself, which can disturb the gut's natural bacteria balance.

Probiotics are live microorganisms that provide health benefits when taken in adequate amounts, while synbiotics are a combination of probiotics and prebiotics (substances that promote the growth of beneficial bacteria). The goal of this study is to explore whether supplementing ESRD patients with probiotics or synbiotics can improve their nutritional health, including aspects like body mass index (BMI), skin fold thickness, and protein metabolism.

The study will involve 60 patients from a hemodialysis center in Mansoura, Egypt. Patients will be randomly assigned to one of three groups: one group will receive probiotics, another will receive synbiotics, and the third group will act as a control (no treatment). The study will evaluate changes in nutritional markers and other health parameters before and after six months of supplementation.

This study hopes to provide insights into new, cost-effective interventions for improving the health of patients undergoing long-term dialysis treatment by addressing the question of whether these supplements can improve the nutritional status of hemodialysis patients.

DETAILED DESCRIPTION:
This randomized controlled trial is designed to assess the effects of probiotic and synbiotic supplementation on the nutritional status of patients with end-stage kidney disease (ESRD) undergoing hemodialysis. Patients with ESRD face significant health challenges, including malnutrition, inflammation, and gut dysbiosis (an imbalance in gut bacteria), which contribute to poor health outcomes and reduced quality of life. These complications are exacerbated by the impact of the hemodialysis process, medications, and dietary restrictions commonly imposed on patients.

Probiotics are live microorganisms that provide health benefits when consumed in adequate amounts. In contrast, synbiotics combine probiotics with prebiotics, which are compounds that selectively stimulate the growth and activity of beneficial gut bacteria. The hypothesis of this study is that both probiotics and synbiotics will improve the nutritional status of hemodialysis patients by enhancing gut microbiota balance, reducing inflammation, and supporting better nutrient absorption.

Study Design: This study will be conducted at the Urology and Nephrology Center in Mansoura, Egypt. A total of 60 patients on regular hemodialysis will be randomly assigned to one of three groups:

Control group (20 patients) - No intervention. Probiotic group (20 patients) - Receives daily probiotic supplementation (Lactogemikan from Pescado Company).

Synbiotic group (20 patients) - Receives daily synbiotic supplementation (Lactogemikan plus prebiotic fiber from oats).

Each group will receive supplementation for a duration of 6 months. The primary goal is to assess the effects of these interventions on the patients' nutritional status, including the monitoring of body mass index (BMI), skin fold thickness, protein catabolic rate (PCR), and subjective global assessment (SGA) of their nutritional health. Additionally, secondary outcomes will include laboratory assessments of serum albumin, cholesterol, and fasting blood glucose.

Methodology: The patients' nutritional parameters will be measured at the start of the study and again after 6 months of supplementation. To assess dialysis adequacy, parameters like the urea reduction ratio and Kt/V (a measure of dialysis efficiency) will be recorded before and after supplementation. These assessments will provide insights into whether probiotics and synbiotics can improve both nutritional markers and dialysis outcomes.

The data will be analyzed using statistical methods including one-way ANOVA, Pearson's and Spearman's correlation, and t-tests to determine the effectiveness of each intervention compared to the control group. The study will ensure the safety and well-being of all participants by monitoring for any adverse effects throughout the trial.

Ethical Considerations: The study will adhere to ethical standards, with approval from the Medical Research Ethics Committee of Mansoura Faculty of Medicine. Informed consent will be obtained from all participants, and their privacy and confidentiality will be maintained throughout the study.

Statistical Analysis: Data will be analyzed using SPSS software (version 26.0). Qualitative data will be presented as counts and percentages, while quantitative data will be presented as means ± standard deviations or medians and interquartile ranges depending on data distribution. Statistical significance will be set at a p-value of ≤ 0.05.

Conclusion: The results of this study will help determine whether probiotics or synbiotics can be used as an effective nutritional intervention for hemodialysis patients. By addressing gut microbiota imbalances and promoting better nutritional health, probiotics or synbiotics could potentially improve patient outcomes and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with End-Stage Renal Disease (ESRD) on regular hemodialysis (3 times per week).
* Age 18 years or older.
* Not prepared for kidney transplantation for more than 1 year.
* Able and willing to provide written informed consent to participate in the study.

Exclusion Criteria:

* Patients who are actively preparing for kidney transplantation.
* Pregnant or breastfeeding women.
* Patients with active malignancy or undergoing cancer treatment.
* Patients with known structural gastrointestinal (GI) disease (e.g., inflammatory bowel disease, severe gastrointestinal motility disorders).
* Patients who have severe infections or other severe conditions that might interfere with the study's assessments.
* Patients with known allergies to probiotics or synbiotics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2025-10-15 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in Body Mass Index (BMI) after 6 Months of Probiotic and Synbiotic Supplementation in Hemodialysis Patients | BMI will be assessed at baseline (before intervention) and at 6 months (after completing the 6-month supplementation period).
  The primary outcome measure will assess the change in Body Mass Index (BMI) as a marker of nutritional status in hemodialysis patients who receive probiotic or synbiotic supplementation. BMI will be measured using standard weight and height measurements at baseline (before supplementation) and at 6 months. A change in BMI will be used to evaluate the overall effect of these interventions on the patients' nutritional status.

SECONDARY OUTCOMES:
Change from Baseline in Serum RAGE Levels after 6 Months of Probiotic and Synbiotic Supplementation in Hemodialysis Patients | Serum RAGE levels will be assessed at baseline (before intervention) and at 6 months (after completing the 6-month supplementation period).
  The secondary outcome measure will assess the change in serum RAGE (Receptor for Advanced Glycation End-products) levels as a marker of oxidative stress and inflammation in hemodialysis patients who receive probiotic or synbiotic supplementation. Serum samples will be collected at baseline (before supplementation) and at 6 months to measure RAGE levels. Changes in RAGE levels will be used to assess the impact of the interventions on oxidative stress and inflammatory markers in these patients.
  RAGE: Elevated levels of RAGE are associated with increased oxidative stress and inflammation, which are common complications in patients with ESRD undergoing hemodialysis.
Change from Baseline in Serum Leptin Levels after 6 Months of Probiotic and Synbiotic Supplementation in Hemodialysis Patients | Serum leptin levels will be assessed at baseline (before intervention) and at 6 months (after completing the 6-month supplementation period).
  This secondary outcome will assess the change in serum leptin levels as a marker of adiposity and metabolic health in hemodialysis patients receiving probiotic or synbiotic supplementation. Serum samples will be collected at baseline (before supplementation) and at 6 months to measure leptin levels. Changes in leptin levels will help determine the impact of the interventions on nutritional status and metabolic dysfunction in these patients.
  Leptin: Leptin is a hormone produced by adipose tissue, and its levels are typically associated with body fat mass and energy balance.

IPD SHARING:
Plan to Share IPD: Undecided
The decision on whether to share individual participant data (IPD) will be determined after the study is completed and the results are published. Factors such as participant consent, data privacy concerns, and the requirements of relevant journals and ethical guidelines will be considered before making a final decision.

REFERENCES:
- [Background] Simoes-Silva L, Araujo R, Pestana M, Soares-Silva I, Sampaio-Maia B. The microbiome in chronic kidney disease patients undergoing hemodialysis and peritoneal dialysis. Pharmacol Res. 2018 Apr;130:143-151. doi: 10.1016/j.phrs.2018.02.011. Epub 2018 Feb 11. PMID 29444477
- [Background] Nguyen TTU, Kim HW, Kim W. Effects of Probiotics, Prebiotics, and Synbiotics on Uremic Toxins, Inflammation, and Oxidative Stress in Hemodialysis Patients: A Systematic Review and Meta-Analysis of Randomized Controlled Trials. J Clin Med. 2021 Sep 28;10(19):4456. doi: 10.3390/jcm10194456. PMID 34640474
- [Background] Liu S, Liu H, Chen L, Liang SS, Shi K, Meng W, Xue J, He Q, Jiang H. Effect of probiotics on the intestinal microbiota of hemodialysis patients: a randomized trial. Eur J Nutr. 2020 Dec;59(8):3755-3766. doi: 10.1007/s00394-020-02207-2. Epub 2020 Feb 28. PMID 32112136
- [Background] Ley RE, Turnbaugh PJ, Klein S, Gordon JI. Microbial ecology: human gut microbes associated with obesity. Nature. 2006 Dec 21;444(7122):1022-3. doi: 10.1038/4441022a. PMID 17183309